CLINICAL TRIAL: NCT00874952
Title: Regional Observation of the Metabolic Syndrome
Acronym: ORSA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Raffaele Sabia/MC MD, AstraZeneca
Other Study IDs: NIS-CIT-DUM-2007/1
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Lipids; Waist Circumference; HDL; hypertension
MeSH Terms: conditions — Metabolic Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study, is to assess the prevalence of metabolic syndrome in Italy on a regional basis, defined according to National Cholesterol Education Program/Adult Treatment Panel III (NCEP/ATPIII) guidelines criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Laboratory analysis (lipidic profile and glycemia) performed in the last year

Exclusion Criteria:

* Subjects with serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's successful participation in the study
* Pregnancy or breast feeding
* Patients enrolled in clinical studies which the aim is to evaluate the efficacy and/or tolerability of anti-hypertensive and/or lipid lowering drugs

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome in primary care population | At visit
Concomitant presence of other cardiovascular (CV) risk factors. | At visit

CONTACTS AND LOCATIONS:
Overall Officials: Mario Mangrella, Study Chair — AstraZeneca S.p.A.; Raffaele Sabia, Study Director — AstraZeneca S.p.A.
Locations (1):
- Research Site, Torino, Italy